CLINICAL TRIAL: NCT02826564
Title: Phase I Trial of Stereotactic Body Radiotherapy With Concurrent Pembrolizumab in Metastatic Urothelial Cancer
Brief Title: Trial of Stereotactic Body Radiotherapy With Concurrent Pembrolizumab in Metastatic Urothelial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/2016/0661 (BC-00197)
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Urothelial Cancer
Keywords: radiotherapy; immunotherapy
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential (Experimental): Stereotactic body radiotherapy prior to pembrolizumab treatment
  Interventions: Drug: pembrolizumab
- Concurrent (Experimental): Stereotactic body radiotherapy concurrent with pembrolizumab treatment
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab
  Other Names: MK-3475

SUMMARY:
The goal of the proposed research project is to assess the safety (dose limiting toxicity, DLT) of the combination of pembrolizumab and high-dose stereotactic body radiotherapy (SBRT) in patients with metastatic urothelial cancer. Both the SBRT dose and pembrolizumab dose will be fixed, but the timing of the combination will be varied. Secondary objectives include response rates, local control, progression-free survival (PFS) and overall survival (OS). Exploratory endpoints include immunologic responses and response rates in PD-L1- TIL- tumors. The combination sequence with the most promising response rates and the best safety profile will be selected to continue in a Phase II trial.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Have measurable disease based on RECIST 1.1.
4. Have had any prior treatment more than 2 weeks prior to study day 1, treatment naïve patients are allowed
5. Histologically confirmed diagnosis of urothelial carcinoma
6. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
7. Have a performance status of 0 or 1 on the ECOG Performance Scale.
8. Demonstrate adequate organ function, all screening labs should be performed within 10 days before treatment initiation.

   (Adequate organ function: Absolute neutrophil count (ANC) ≥1,500 /mcL, Platelets ≥100,000 / mcL, Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment), Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN, Serum total bilirubin ≤ 1.5 X ULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN, AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases, Albumin >2.5 mg/dL, International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy (as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants a Creatinine clearance should be calculated per institutional standard)
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has had radiotherapy interfering with SBRT.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has a known history of active TB (Bacillus Tuberculosis)
5. Hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Selection of the sequence arm with a DLT < 20% based on the incidence of treatment-related adverse events | 12 weeks post-radiotherapy
  Toxicities will be considered as DLT if occurring between the start of SBRT and 12 weeks after completion of SBRT. DLT will be assessed using the Common Terminology Criteria for Adverse Events.

SECONDARY OUTCOMES:
Tumor response | 12 weeks
  Response rate of non-irradiated lesions will be evaluated as per RECIST v1.1 and per immune related response criteria (irRC) (Wolchok et al Clinical Cancer Research 2009)
Immunologic response in peripheral blood | 12 weeks
  Immunologic responses will be assessed using peripheral blood samples, analyzed with FACS phenotyping, functional testing and ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Result] Sundahl N, Vandekerkhove G, Decaestecker K, Meireson A, De Visschere P, Fonteyne V, De Maeseneer D, Reynders D, Goetghebeur E, Van Dorpe J, Verbeke S, Annala M, Brochez L, Van der Eecken K, Wyatt AW, Rottey S, Ost P. Randomized Phase 1 Trial of Pembrolizumab with Sequential Versus Concomitant Stereotactic Body Radiotherapy in Metastatic Urothelial Carcinoma. Eur Urol. 2019 May;75(5):707-711. doi: 10.1016/j.eururo.2019.01.009. Epub 2019 Jan 19. PMID 30665814
- [Result] Sundahl N, De Wolf K, Rottey S, Decaestecker K, De Maeseneer D, Meireson A, Goetghebeur E, Fonteyne V, Verbeke S, De Visschere P, Reynders D, Van Gele M, Brochez L, Ost P. A phase I/II trial of fixed-dose stereotactic body radiotherapy with sequential or concurrent pembrolizumab in metastatic urothelial carcinoma: evaluation of safety and clinical and immunologic response. J Transl Med. 2017 Jun 29;15(1):150. doi: 10.1186/s12967-017-1251-3. PMID 28662677
- See also: Article — https://translational-medicine.biomedcentral.com/counter/pdf/10.1186/s12967-017-1251-3.pdf